CLINICAL TRIAL: NCT00005358
Title: Thrombogenic Factors and Recurrent Coronary Events
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4245; R01HL048259 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Myocardial Infarction; Thrombosis; Death, Sudden, Cardiac
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Myocardial Infarction; Thrombosis; Death, Sudden, Cardiac

SUMMARY:
To determine if selected circulating blood factors that reflect enhanced thrombogenesis are associated with an increased incidence of recurrent coronary events, including cardiac death or non-fatal myocardial infarction.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

In this multicenter, collaborative, prospective study, patients hospitalized with a myocardial infarction were enrolled from ten geographically dispersed centers. Five thrombogenic- related blood factors were quantitated, and formed the centerpiece of this study: 1) lipoprotein(a) [Lp(a)] - a quantitative genetic factor that contains apolipoprotein B, has a structural homology to plasminogen, interferes with intrinsic thrombolytic activity, and represents a crossover link in the thrombogenesis/atherogenesis hypothesis; 2) soluble fibrin - a system indicator of coagulation activity in the ongoing conversion of fibrinogen to insoluble fibrin strands; 3) plasminogen activator inhibitor-1 (PAI-1) - an important regulator of the fibrinolytic system, it interferes with intrinsic t-PA activity; 4) coagulation Factor VII -high levels lead to increased thrombogenesis and have been associated with an increased risk of ischemic heart disease; and- 5) von Willebrand factor - it binds to platelet glycoproteins, contributes to local thrombus formation, and it is elevated in patients at increased risk of coronary thrombosis.

The primary analysis utilized a time-dependent survivors hip model (Cox regression) to determine the presence or absence of an association between one or more of these factors and subsequent thrombotic-related coronary events. Secondary objectives included: 1) to determine if there was a statistical association between the thrombogenic factors and conventional hematologic/lipid parameters, and to evaluate their interactions regarding coronary events; and 2) to determine if thrombogenic factors had uniform effects on coronary event rates across various subgroups.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1994-04; Study Completion 1999-03

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Moss — University of Rochester

REFERENCES:
- [Background] Marder VJ, Zareba W, Horan JT, Moss AJ, Kanouse JJ. Automated latex agglutination and ELISA testing yield equivalent D-dimer results in patients with recent myocardial infarction. THROMBO Research Investigators. Thromb Haemost. 1999 Nov;82(5):1412-6. PMID 10595629
- [Background] Moss AJ, Goldstein RE, Marder VJ, Sparks CE, Oakes D, Greenberg H, Weiss HJ, Zareba W, Brown MW, Liang CS, Lichstein E, Little WC, Gillespie JA, Van Voorhees L, Krone RJ, Bodenheimer MM, Hochman J, Dwyer EM Jr, Arora R, Marcus FI, Watelet LF, Case RB. Thrombogenic factors and recurrent coronary events. Circulation. 1999 May 18;99(19):2517-22. doi: 10.1161/01.cir.99.19.2517. PMID 10330382